CLINICAL TRIAL: NCT07048717
Title: The Mauritius and Rodrigues Non-Communicable Disease (NCD) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Ministry of Health and Wellness, Mauritius (Unknown); University of Helsinki (Other); Monash University (Other); Imperial College London (Other); Baker Heart and Diabetes Institute (Other)
Responsible Party: Principal Investigator, Stefan Soderberg, Professor, consultant, Umeå University
Other Study IDs: 2023-07199-01
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diabete Mellitus; Cardiovascular Disease Risk Factor; Ischemic Cardiovascular Disease; Hypertension; Obesity &Amp; Overweight
Keywords: Epidemiology; Cross-sectional studies; Prevalence; Incidence; Diabetes mellitus; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Obesity; Overweight; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples Without DNA — Plasma samples from the last surveys (2021 an 2022) are stored locally in Mauritius
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Randomly selected population-based subjects from the population (Mauritius): Seven cross-sectional studies were performed between 1987 and 2021 on mainland Mauritius
- Randomly selected population-based subjects from the population (Rodrigues): In parallell, six cross-sectional studies were performed between 1992 and 2022 on Rodrigues

SUMMARY:
Mauritius is located in the southern Indian Ocean with a population of 1.3 million in 2023. Mauritius is a multiethnic nation with 68% South Asian, 27% African (Creole), 3% Chinese and 2% Franco Mauritians.

Seven population-based cross-sectional surveys using standardised protocols were conducted between 1987 and 2021). The participation rate has been over 85% in each survey.

At each survey, participants were interviewed about living conditions, lifestyle and health, and anthropometry and blood pressure were measured. Biochemistry including lipids and an oral glucose tolerance test (OGTT) were performed Electrocardiograms (ECG) were recorded in participants aged 35 years and older. Previous participants were followed up in 2007 and 92% were successfully traced.

Studies with identical methodology have been performed on the neighbouring island Rodrigues where the majority of the population are Creoles.

DETAILED DESCRIPTION:
Mauritius and Rodrigues are islands in the south-eastern part of the Indian Ocean. Major changes in lifestyle have been seen during the last fifty years, including less physical activity and introduction of a westernised diet. In parallel, the disease panorama has changed from high infant mortality and infectious diseases to lifestyle-related diseases such as cardiovascular disease and type 2 diabetes.

The population in Mauritius are descendants to immigrants from South Asia, Africa and China, i.e., approximately 60% of the world population are represented. Mauritius is probably the only developing country that has followed the development of non-communicable diseases (NCD) and associated risk factors over a long time-period and continues to do so.

In the mid-eighties, the Mauritian government initiated a study on the prevalence of type 2 diabetes and cardiovascular disease, in collaboration with WHO and international experts. Altogether seven population-based surveys have been performed between 1987 and 2021, and approximately 39 000 (!) examinations have been recorded. The intention is to repeat the survey every fifth year.

The ethnicities of the participants have been 71% South Asians (India/Pakistan), 24% Creoles (Africa) and 5% Chinese, which reflects well the ethnical distribution of the population. Previous participants were followed up in 2007 and 92% were successfully traced. Studies have also been performed on the neighbouring island Rodrigues where the majority of the population are Creoles. During the follow-up survey in 2010, 97% of the 9 700 participants were traced.

At each survey, information was given and an individual consent form was signed. See attached the local (in Mauritius) ethical approval and consent form from the Mauritius survey 2021.

At each survey, participants were interviewed about living conditions, lifestyle and health, and anthropometry and blood pressure were measured. Biochemistry including lipids and an oral glucose tolerance test (OGTT) were performed Altogether approximately 28 000 electrocardiograms (ECG) were recorded in participants aged 35 years and older, all of which have been coded in Kaunas, Lithuania for signs of ischemic heart disease (Minnesota criteria) and myocardial hypertrophy.

The Mauritius NCD study was initially administrated by the International Diabetes Institute in Melbourne, Australia under the leadership of Professor Paul Zimmet together with Professor Jaakko Tuomilehto (Finland) and Professor George Alberti (United Kingdom). Today, the study is administrated and financed by the Ministry of health in Mauritius under the leadership of Doctor Sudhir Kowlessur.

Professor Stefan Söderberg at the Department of Public Health and Clinical Medicine, Umeå University, Sweden was introduced to the Mauritius NCD study during his postdoc (2001-2002) in Professor Zimmet's research team at IDI in Melbourne. Söderberg has since then continued to assist in the performance of the surveys and to analyse data. Today, Umeå university and the Department of Public Health and Clinical medicine have been granted the privilege to curate and analyse data generated in the Mauritius and Rodrigues NCD study.

Each survey has been evaluated and approved by the local ethics committee in Mauritius (see attached the approval from 2021). Analysing data in Sweden has been approved by the Swedish Ethical Authority (2023-07199-01).

ELIGIBILITY:
In short:

Inclusion

* Men and women
* Randomly selected population-based samples (details see below)
* Target age from 25 to 74 years Exclusion
* Not living in the study area
* Age outside the age-range

In detail:

Inclusion Criteria In 1987, 10 randomly selected (with probability proportional to size) population clusters and a purposely selected area of Chinatown in the capital, Port Louis, were surveyed (age range 25-74), and all eligible residents were invited to participate.2 In 1992 and 1998, the same clusters were resurveyed as well as an additional three clusters selected to assess if trends in disease and risk factor distribution observed in the study cohort also occurred in independent clusters (age range 25 years and older). In 1998, the Chinatown cluster was not surveyed. Altogether, 9,559 individuals participated in the first three surveys and 60% of participants took part in more than one survey.

In 2004, a new study was performed, with similar methodology. In 2009, nine index clusters were chosen with one randomly selected from each of the nine districts in Mauritius. Then, two neighbouring clusters were chosen surrounding the index cluster to form a "super cluster." From this super cluster, one in three households was randomly selected and one adult per household was invited to participate.5 The same methodology was used in 2015 and in 2021 with new randomly chosen clusters forming "super cluster" as in 2009. In addition, a random sample from the 1998 survey was invited for a resurvey in 2015.

Participation rate has been over 85% in each survey. No sampling weights were used.

Same methodology was used in Rodrigues.

Exclusion Criteria Outside age-range and not being randomly selected.

Ages: 25 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random samples from the Mauritian (including Rodrigues) aged 25 to 74 years
Sampling Method: Probability Sample
Enrollment: 39082 (Actual)
Dates: Start 1987-04-05 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | Up to 20 years from the baseline survey
  According to household interviews, death certificates from central registers at Ministry of Health and Wellness.
  1. Household interviews: "Is the participant alive? If dead, do you have a copy of the death certificate? When did the participant die?"
  2. Central registers: Vital status, if dead, date and cause of death from death certificates"
  Combining 1 and 2 will give date and cause of death.
  Absolute numbers and mortality rates will be reported for all and in subgroups i.e. sex, age-strata, ethnicity.

SECONDARY OUTCOMES:
Diabetes Mellitus | Up to 20 years from the baseline survey
  Determined according to WHO criteria. i.e. data from oral glucose tolerance tests and questionnaires (glucose-lowering medication).
  1. A 75-g oral glucose-tolerance test is used on all non-pregnant participants, except those taking insulin or oral hypoglycaemic drugs, was performed after an overnight fast, and plasma glucose (mmol/L) are measured before the test and after two hours.
  2. The questionnaire includes the question: "Do you take glucose-lowering medication, insulin or tablets, yes/no".
  The participant has diabetes if fasting glucose ≥ 7.0 mmol/ and/or two-hour glucose ≥ 11.1 mmol/L and/or answer yes to taking glucose lowering medication, and prediabetes if fasting glucose ≥ 6.1 and < 7.0 mmol/L and/or two-hour glucose ≥ 7.8 and < 11.1 mmol/L.
  Numbers and age-standardised incidence and prevalence of prediabetes and diabetes will be reported for all and in subgroups.
Cardiovascular disease (CVD) | Up to 20 years from the baseline survey
  Determined by analysis of serial ECG recordings, data from official registers and questionnaires.
  ECGs and signs of coronary heart disease (CHD) according to the Minnesota Code (MC) classification. Probable CHD (MC: 1-1 to 1-2 (large Q and QS)) and possible (CHD) (MC: 1-3 (small Q and QS), 4-1 to 4-4 (ST depression), 5-1 to 5-3 (T wave inversion and flat) and 7-1 (left bundle branch block)). Probable CHD will be interpreted as previous myocardial infarction (MI).
  From central registers: Date and related ICD 10 codes for hospital admissions. ICD codes I21-23 will be interpreted as MI, and I60-61 and I63-64 as stroke.
  Survey: Affirmative answer to any of these questions: Do you have angina, myocardial infarction (including by-pass surgery and PCI), and/or stroke" will be labelled as previous CVD.
  CVD is present if probable CHD and/or ICD codes found for MI or stroke and/or affirmative answer to surve questions.
Hypertension | Up to 20 years from the baseline survey
  Blood pressure (BP) is measured using an automated BP monitor (Omron Digital Auto Blood Pressure Monitor).
  The questionnaire includes the question: "Do you take BP lowering medication, yes/no".
  Hypertension is defined as a systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg, and/or answer "yes" to the use of BP lowering drugs.
  Numbers and age-standardised incidence and prevalence of hypertension will be reported for all and in subgroups.
Obesity | Up to 20 years from the baseline survey
  Height (in meter, m) and weight (in kilogram, kg) will be measured in light clothing without shoes.
  Waist circumference (in centimeter, cm) is measured as the circumference at the mid-point between the iliac crest and the lower margin of the ribs. Hip circumference (in centimeter, cm) is taken as the horizontal measure around the pelvis at the point of maximal protrusion of the buttocks.
  Waist and hip circumference are measured twice, and the mean will be calculated.
  Body mass index (BMI) is calculated as weight divided by height squared (kg/m2), and waist to hip ratio (WHR) as waist circumference (cm) divided by hip circumference (cm).
  Obesity is defined according to BMI as ≥ 30 kg/m2, and central obesity according to waist circumference using ethnic-specific cut-offs.
  Numbers and age-standardised incidence and prevalence of obesity and central obesity will be reported for all and in subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Zimmet, Professor, Principal Investigator — Monash University; George Alberti, Professor, Principal Investigator — Imperial College, London, UK; Jaakko Tuomilehto, Professor, Principal Investigator — Helsinki University, Helsinki, Finland
Locations (1):
- Port Louis, Mauritius

IPD SHARING:
Plan to Share IPD: Yes
If you would like to use the data from the Mauritius study, you should contact the Section of Biobank and Registry Support (BRS) at Umeå University, Sweden for discussion: info.brs@umu.se.
  Before sharing of data, the application will be evaluated by senior researchers within the network. Ethical approval must be obtained.
Supporting Information: Study Protocol
Time Frame: Available now
Access Criteria: Reasonable request approved by senior researchers within the study group, plus obtained ethical approval.
URL: https://www.umu.se/en/research/groups/the-mauritius-study/

REFERENCES:
- [Result] Soderberg S, Taki H, Kowlessur S, Shaw JE, Magliano DJ, Tamosiunas A, Alberti G, Zimmet P, Tuomilehto J. Trends in the prevalence of cardiovascular disease, defined as ECG abnormalities and/or self-reported events, in Mauritius between 1987 and 2021: analysis of data from seven large population-based surveys. BMJ Open. 2025 Jun 16;15(6):e087693. doi: 10.1136/bmjopen-2024-087693. PMID 40523792
- See also: Description of the Mauritian/Rodrigues NCD survey at Umeå University, Sweden — https://www.umu.se/en/research/groups/the-mauritius-study/
- Available data/document: General information about the study plus information about application for data — https://www.umu.se/en/research/groups/the-mauritius-study/

DOCUMENTS (1):
  • Informed Consent Form (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT07048717/ICF_000.pdf